CLINICAL TRIAL: NCT03182010
Title: Ultrasound Evaluation of Cesarean Scar After Uterotomy Closure With Barbed and Conventional Sutures ; a Randomized Controlled Study
Brief Title: Ultrasound Evaluation of Cesarean Scar After Uterotomy Closure With Barbed and Conventional Sutures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Usama M Fouda, Prof., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Barbed sutures/Cesarean scar
Record Dates: First submitted 2017-06-07; First posted 2017-06-09 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Cesarean Section Scar
Keywords: Cesarean section scar, Barbed suture, Conventional suture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cesarean section incision closure using barbed sutures (Experimental): Cesarean section incision is closed using barbed sutures
  Interventions: Device: Cesarean section incision closure using barbed sutures
- Cesarean section incision closure using conventional sutures (Active Comparator): Cesarean section incision is closed using conventional sutures
  Interventions: Device: Cesarean section incision closure using conventional sutures

INTERVENTIONS:
Device: Cesarean section incision closure using barbed sutures — Cesarean section incision will be closed using a 24-cm × 24-cm 0 polydioxanone double-armed suture on a 26-mm half-circle reverse cutting needle( STRATAFIX™ Spiral PDO Knotless Tissue Control Device, Ethicon Inc , Somerville, NJ, USA ).Ultrasound examination will be performed 6 months after the operation to measure the residual myometrial thickness and the scar depth.
  Arms: Cesarean section incision closure using barbed sutures
Device: Cesarean section incision closure using conventional sutures — Cesarean section incision will be closed using 1-0 polyglactin 910 suture(VICRYL™.; Ethicon Inc, Sommerville, NJ) .Ultrasound examination will be performed 6 months after the operation to measure the residual myometrial thickness and the scar depth.
  Arms: Cesarean section incision closure using conventional sutures

SUMMARY:
The aim of this randomized control trial is to compare the residual myometrial thickness and the depth of cesarean section scar defect after uterine incision closure with barbed or conventional sutures.

DETAILED DESCRIPTION:
The aim of this randomized control trial is to compare the residual myometrial thickness and the depth of cesarean section scar defect after uterine incision closure with barbed or conventional sutures. Primigravida patients undergoing transverse lower segment cesarean section will be included in the study.Cesarean section incision will be closed with double layers of continuous barbed or conventional sutures. Ultrasound examination will be performed 6 months after the operation to measure the residual myometrial thickness and the scar depth.

ELIGIBILITY:
Inclusion Criteria:

* Primigravida patients undergoing transverse lower segment cesarean section

Exclusion Criteria:

* Previous laparotomies
* Postoperative fever
* Patients with preterm pregnancies or in labor

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 110 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Residual myometrial thickness | Six months after cesarean section
  Thickness of myometrium under the niche

SECONDARY OUTCOMES:
Scar depth | Six months after cesarean section

CONTACTS AND LOCATIONS:
Overall Officials: Usama M Fouda, Prof., Study Chair — Cairo University; Mohamed Zayed, Prof., Principal Investigator — Cairo University
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No